CLINICAL TRIAL: NCT07383506
Title: A Study of a Mutant-Selective Inhibitor, CGT6297, in Patients With Advanced Solid Tumors Harboring PIK3CA Mutations
Brief Title: A Study of Mutant Selective-Inhibitor (CGT6297), in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CGT6297-25-101
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: PIK3CA Mutations; Advanced Solid Tumors, Adult; Endometrial Cancer; HR Positive/HER-2 Negative Breast Cancer; HER2-low Breast Cancer
Keywords: HER2; PI3K; Mutant-Selective Inhibitor; Advanced solid tumors; PIK3CA Mutations; PIK3CA SNVs; Endometrial Cancer; Breast Cancer; HR+/HER2 Negative breast cancer; HR+/HER2 (-) breast cancer; HR+/HER2 low breast cancer; PI3KCA Genetic Alterations; PI3KCA Point Mutations; PI3KCA Gene Short Variants; PI3KCA active alteration; HER2-low Breast Cancer; Phase 1a/1b
MeSH Terms: conditions — Endometrial Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1, Part A evaluating multiple ascending doses Phase 1b, evaluation of Part A selected doses in 3 cohorts defined by tumor type including a randomized dose optimization design (Part B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Part 1a: Dose Escalation of Multiple doses of CGT6297 for oral administration
  Interventions: Drug: CGT6297
- Signal Seeking (Experimental): Phase 1b: Participants will receive CGT6297 at a dose level selected based on data from Phase 1a
  Interventions: Drug: CGT6297

INTERVENTIONS:
Drug: CGT6297 — CGT6297 Daily Oral Administration

SUMMARY:
This is a Phase 1, two-part, open-label, nonrandomized, dose-escalation and signal-seeking study of CGT6297, evaluating the safety, tolerability, PK, pharmacodynamic (what the drug does to the body), and antitumor activity of CGT6297 in adult participants with advanced solid tumors harboring PIK3CA mutations

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced solid tumor harboring oncogenic PIK3CA mutations in blood and/or tumor:

   1. Phase 1b Cohort 1, participants must have PIK3CA endometrial cancer
   2. Phase 1b Cohort 2, participants must have HR-positive/HER2-negative or HER2-low breast cancer (immunohistochemistry [IHC] and in-situ hybridization results must meet ASCO-College of American Pathology guidelines for breast cancer or criteria)
   3. Phase 1b Cohort 3 will allow all solid tumors that do not meet criteria for Phase 1b Cohorts 1 or 2, including head and neck cancers, other gynecological cancers, colorectal cancers harboring PIK3CA mutations
2. Meet prior treatment requirement of:

   1. Phase 1a: previously treated with and refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.
   2. Phase 1b: previously treated with or considered not appropriate for SOC first-line treatment for their condition
3. Have at least one measurable lesion according to RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
5. Have clinically acceptable local laboratory screening results (clinical chemistry and hematology) within certain limits
6. Resolution of acute toxicities from prior anticancer therapy to ≤Grade 1 (or baseline), including resolution of clinically significant laboratory abnormalities (other than parameters specified in screening testing as outlined below), as determined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCICTCAE) v5.0.
7. Have an ejection fraction ≥50%

Exclusion Criteria:

1. Received small molecule chemotherapy or anticancer therapies or radiotherapy within certain timeframes before first dose of study drug.
2. Major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of study drug
3. Treatment with radiotherapy ≤2 weeks before the first dose of study drug.
4. Clinically significant cardiac disease
5. Ongoing or planned long-term (≥4 consecutive weeks) treatment with glucocorticoid steroids at greater than physiologic dosing (defined as equivalent to >20 mg/day prednisone)
6. Diagnosis of diabetes mellitus type 1 or uncontrolled diabetes mellitus type 2 (defined as fasting glucose ≥140 mg/dL and HbA1c ≥7.0%; antihyperglycemic medical management permitted with the exception of insulin)
7. Previous molecular testing (NGS or PCR) showed tumor with the following mutations: mutations/deletions in PTEN or activating mutations in AKT, HRAS/KRAS/NRAS, EGFR, and BRAF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) [Phase 1a] | Approximately 12 months
  Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) and AEs leading to dose modifications and dose limiting toxicities (DLTs) to determine the maximum tolerated dose (MTD) or the maximum evaluated dose (MED) of CGT6297 in participants with advanced solid tumors harboring PIK3CA mutations
Overall Response Rate [Phase 1b] | Approximately 8 months
  Overall Response Rate (ORR), as determined by CR + PR based on Investigator assessment using RECIST v1.1

SECONDARY OUTCOMES:
Incidence and grade of Adverse Events (AEs) and Serious Adverse Events (SAEs) [Phase 1b] | Approximately 12 months
  * Incidence and grade of Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs leading to dose modification
  * Changes from baseline in key laboratory results and electrocardiogram (ECG) parameters
Pharmacokinetics (Part 1a) | Approximately 28 days
  Area under the concentration-time curve (AUC) in participants with advanced solid tumors harboring PI3K mutations
Pharmacokinetics (Part 1a) | Approximately 28 days
  Maximum observed concentration (Cmax) in participants with advanced solid tumors harboring PI3K mutations
Pharmacokinetics (Part 1a) | Approximately 28 days
  Observed concentration at predose (Ctrough) in participants with advanced solid tumors harboring PI3K mutations
Pharmacokinetics (Part 1a) | Approximately 28 days
  Time to maximum concentration (Tmax) in participants with advanced solid tumors harboring PI3K mutations
Disease Response (Part 1b) | Approximately 8 months
  Objective response rate (ORR), determined by confirmed (CR) + (PR) based on Investigator assessment using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Disease Response (Part 1b) | Approximately 28 days
  Disease control rate (DCR), as determined by confirmed CR + PR + stable disease (SD) based on Investigator assessment using RECIST v1.1

IPD SHARING:
Plan to Share IPD: No